CLINICAL TRIAL: NCT02127710
Title: A Phase II Trial to Evaluate the Efficacy of AZD6094 (HMPL-504) in Patients With Papillary Renal Cell Carcinoma (PRCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5082C00002; GU 111 (Other: Sarah Cannon Research Institute (SCRI))
Record Dates: First submitted 2014-04-23; First posted 2014-05-01 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Papillary Renal Cell Cancer
Keywords: AZD6094; Savolitinib; Papillary Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD6094 600 mg daily continuously (Experimental): All patients entering the study will take AZD6094 600 mg by mouth (PO) once daily (QD). Treatment will be given continuously.
  Interventions: Drug: AZD6094

INTERVENTIONS:
Drug: AZD6094 — AZD6094 is a potent and selective small molecule mesenchymal epithelial transition (c-MET) kinase inhibitor.
  Other Names: Savolitinib; HMPL - 504

SUMMARY:
This is an open-label, single-arm, multicentre, global, phase II study designed to evaluate the efficacy and safety of AZD6094 in patients with papillary renal cell carcinoma (PRCC) who are treatment naïve or previously treated.

An independent central pathology review of tumour samples will be used to confirm the diagnosis of PRCC of all patients enrolling. However, locally available pathology results confirming PRCC will be allowed for timely study entry.

DETAILED DESCRIPTION:
The study will comprise two stages. In Stage 1 approximately 20 patients will be enrolled. This group is considered sufficient to provide preliminary assessment of the anti-tumour activity of AZD6094 in the form of non-binding futility analysis.

If ≤ 2 tumour responses are observed in the first 20 evaluable patients termination of the study will be considered taking into account the relevant molecular profile of the patients and additional information from related studies in the drug development programme.

All patients entering the study will take AZD6094 600 mg by mouth (PO) once daily (QD). Treatment will be given continuously.

Following the baseline assessment, efficacy will be assessed by objective tumour assessments every 6 weeks (±7 days), for the first 12 months and every 12 weeks thereafter until objective disease progression as defined by RECIST v1.1 There will be a data cut-off after all patients have completed at least 12 weeks of treatment with AZD6094 or withdrawn. The database will be locked and data analysis will be performed on this dataset.

Any patients still receiving study drug at the time of data cut-off will be able to continue to receive AZD6094 while deriving clinical benefit. Such patients will continue to be monitored for the occurrence of serious adverse events up to 28 days after the last dose of AZD6094.

After database lock (DBL) tumour assessments will be performed every 12 weeks (±7 days) until objective disease progression as defined by RECIST v1.1.

Patients discontinuing treatment due to documented disease progression will enter a survival follow-up period, where they will be followed for the initiation of subsequent anti-cancer therapies every 3 months until death, loss to follow-up or withdrawal of consent, whichever comes first.

Patients discontinuing treatment prior to documented disease progression will enter a progression-free survival follow-up period where they will continue to have disease assessments every 6 weeks (±7 days) for the first 12 months of follow-up and every 12 weeks thereafter until objective disease progression as defined by RECIST v1.1, death, loss to follow-up or withdrawal of consent, whichever comes first. After DBL, tumour assessments will be performed in the progression free survival patient population every 12 weeks (±7 days) until objective disease progression as defined by RECIST v1.1

ELIGIBILITY:
Inclusion criteria

1. Provision of informed consent prior to any study specific procedures, sampling and analyses.
2. Histologically confirmed PRCC, which is locally advanced or metastatic.
3. Availability of an archival tumor sample or a pre-treatment fresh tumor sample for confirmation of PRCC by a central laboratory and other biomarker
4. Treatment naïve or have failed on previous treatment for PRCC. Previous treatments may include: targeted therapy (i.e. sunitinib, sorafenib, bevacizumab, pazopanib, temsirolimus, and everolimus), traditional immunotherapy (i.e. interferon-a, Interleukin-2), chemotherapy or a combination of chemoimmunotherapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. At least one lesion, not previously irradiated, and not chosen for a biopsy if performed during the screening period that can be accurately measured at baseline and which is suitable for accurate repeated measurements.
7. Adequate hematological function defined as:

   1. Absolute neutrophil count ≥1500/μL
   2. Haemoglobin ≥9 g/dL
   3. Platelets ≥100,000/μL
8. Adequate liver function defined as:

   1. Alanine aminotransferase and aspartate aminotransferase ≤2.5 x the upper limit of normal (ULN)
   2. Total bilirubin ≤1.5 x ULN
9. Adequate renal function defined as glomerular filtration rate ≥ 40 mL/min,
10. Adequate coagulation parameters, defined as International Normalisation Ratio <1.5 x ULN or activated partial thromboplastin time <1.5 x ULN.
11. Patients with known tumor thrombus or deep vein thrombosis are eligible if stable on low molecular weight heparin for ≥4 weeks.
12. Females should be using adequate contraceptive measures should not be breast feeding, and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential
13. Male patients should be willing to use barrier contraception, i.e. condoms.
14. Ability to swallow and retain oral medications.
15. Predicted life expectancy ≥12 weeks.
16. Aged at least 18 years.
17. Willingness and ability to comply with study and follow-up procedures.
18. Ability to understand the nature of this study and give written informed consent.

Exclusion criteria

1. Most recent chemotherapy, immunotherapy, chemo-immunotherapy, or investigational agents <21 days of the first dose of study treatment. Most recent targeted therapy <14 days of the first dose of study treatment.
2. Unresolved toxicities from any prior therapy greater than Common Terminology Criteria for Adverse Events Grade 1 at the time of starting study treatment with the exception of alopecia.
3. Prior or current treatment with a cMet inhibitor
4. Strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4), strong inhibitors of cytochrome P450 1A2 (CYP1A2), or CYP3A4 substrates with a narrow therapeutic range within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort)
5. Wide field radiotherapy (including therapeutic radioisotopes such as strontium-89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy
6. Major surgical procedures ≤28 days of beginning study drug or minor surgical procedures ≤7 days. No waiting is required following port-a-cath placement.
7. Previously untreated brain metastases.
8. Current leptomeningeal metastases or spinal cord compression due to disease.
9. Acute or chronic liver or pancreatic disease.
10. Uncontrolled diabetes mellitus.
11. Gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy
12. Any of the following cardiac diseases currently or within the last 6 months:

    1. Unstable angina pectoris
    2. Congestive heart failure (New York Heart Association ≥ Grade 2)
    3. Acute myocardial infarction
    4. Stroke or transient ischemic attack
13. Inadequately controlled hypertension (i.e., systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg) (patients with values above these levels must have their blood pressure controlled with medication prior to starting treatment).
14. Mean resting correct QT interval (QTc) >470 msec obtained from triplicate electrocardiagrams
15. Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiograms, e.g. complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec.
16. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital or familial long QT syndrome or family history of unexplained sudden death under 40 years of age or any concomitant medications known to prolong QT interval.
17. Currently receiving treatment with therapeutic doses of warfarin sodium. Low molecular weight heparin is allowed.
18. Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
19. Known diagnosis of human immunodeficiency virus, hepatitis B, or hepatitis C.
20. Presence of other active cancers, or history of treatment for invasive cancer ≤5years. Patients with Stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
21. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-04-14 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik-Tobias Arkenau, MD,PhD, Study Chair — Sarah Cannon Research Institute United Kingdom
Locations (21):
- United States (13):
  - Research Site, Birmingham, Alabama
  - Research Site, Duarte, California
  - Research Site, Palo Alto, California
  - Research Site, Fort Myers, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
- Research Site, Barcelona, Spain
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D5082c00002-revised-csp-3_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2609&filename=d5082c00002-revised-csp-3_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 111 patients were enrolled; 109 patients received at least one dose of AZD6094 administered orally (po). Two patients withdrew prior to receiving any study drug. The study was conducted at 23 international sites in the United States, Canada, United Kingdom and Spain.
Pre-assignment Details: All patients were required to provide an archived or fresh tumour sample at enrolment to confirm eligibility, and for performance of the c-MET biomarker analysis. c-MET biomarker results determined the subgroup placement for data analysis as follows: c-MET positive (n=46), c-MET negative (n=47), and c-MET unknown (n=16).
Groups:
- c-MET Positive [600mg AZD6094 po]: All participants tested for the presence of c-MET mutations
- c-MET Negative [600mg AZD6094 po]; c-MET Status Unknown [600mg AZD6094 po]: All participants were tested for the presence of c-MET mutations.
Period: Overall Study
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po]
Started | 46 | 47 | 16
Completed | 46 | 47 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of AZD6094 are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po] | Total
Number analyzed (Participants) | 46 | 47 | 16 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 9 | 59
  >=65 years | 22 | 21 | 7 | 50
Age, Continuous [Median (Full Range); unit: years] | 64 [23 to 87] | 64 [29 to 75] | 61 [37 to 80] | 64 [23 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 7 | 31
  Male | 33 | 36 | 9 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 2 | 14
  Not Hispanic or Latino | 40 | 41 | 14 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status (PS): (0) = Fully active; (1) Restricted in physically strenuous activity; (2) Ambulatory and capable of self-care; (3) Capable of limited self-care; (4) Completely disabled
  Participants
    PS=0 | 19 | 25 | 7 | 51
    PS=1 | 27 | 22 | 9 | 58
    PS=2 | 0 | 0 | 0 | 0
    PS=3 | 0 | 0 | 0 | 0
    PS=4 | 0 | 0 | 0 | 0
PRCC Confirmation from Central Laboratory [Count of Participants; unit: Participants]
  PRCC Not Confirmed | 9 | 7 | 8 | 24
  PRCC Confirmed | 37 | 40 | 8 | 85
Stage Classification [Count of Participants; unit: Participants]
  Low | 1 | 4 | 0 | 5
  Intermediate | 8 | 12 | 4 | 24
  High | 13 | 15 | 3 | 31
  Missing | 24 | 16 | 9 | 49
Renal Cell Classification [Count of Participants; unit: Participants]
  Type I PRCC | 12 | 2 | 2 | 16
  Type II PRCC | 25 | 38 | 6 | 69
  Unclassified PRCC | 7 | 5 | 2 | 14
  Other | 0 | 1 | 1 | 2
  Unknown | 2 | 1 | 5 | 8
MSKCC Risk Group [Count of Participants; unit: Participants] — Risk categories for patients were obtained from the Memorial Sloan Kettering Cancer Center (MSKCC) risk category prognostic model in advanced renal cell cancer, as follows: Favourable risk = 0 risk factors; Intermediate risk = 10 or 2 risk factors; Poor risk = 3 or more risk factors. Risk factors include: Karnofsky performance status < 80%; time from diagnosis to salvage treatment < 1 year; haemoglobin < lower limit of normal (LLN); corrected serum calcium > ULN; and serum lactate dehydrogenase > 1.5 x ULN.
  Participants
    Favourable Risk | 3 | 10 | 2 | 15
    Intermediate Risk | 28 | 14 | 7 | 49
    Poor Risk | 3 | 5 | 2 | 10
    Missing | 12 | 18 | 5 | 35
Weight [Mean (Standard Deviation); unit: kilograms] | 78.42 (20.74) | 85.38 (23.84) | 84.90 (12.55) | 82.37 (21.32)
Weight [Median (Full Range); unit: Kg] | 76.5 [42 to 134] | 83.5 [47 to 160.6] | 87.65 [59.3 to 101.6] | 79.5 [42 to 160.6]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (RECIST Version 1.1)
Description: The primary outcome measure was Objective Response Rate (ORR), defined as the proportion of patients with either a complete response or a partial response by investigator assessment according to Response Evaluation Criteria for Solid Tumours (RECIST) v1.1.
Time Frame: Up to 12 months
Population: ORR was assessed on the efficacy analysis set, consisting of all patients with measurable disease, PRCC confirmed by a central laboratory and have received at least 1 dose of AZD6094 (n = 85).
Measure: Count of Participants; unit: Participants
Groups:
- Efficacy Analysis Set: All patients with measurable disease, PRCC confirmed by central laboratory and received at least 1 dose of study medication
- Safety Analysis Set: All patients who have received at least 1 dose of study medication
Arm/Group | Efficacy Analysis Set | Safety Analysis Set
Number analyzed (Participants) | 85 | 109
Participants
  Complete Response | 0 | 0
  Partial Response | 3 | 8
  Stable Disease >= 5 Weeks | 46 | 59
  Progression | 34 | 40
  Not Evaluable | 2 | 2

2. Primary Outcome: Objective Response Rate (RECIST Version 1.1) Stratified by c-MET Status in Efficacy Analysis Set
Description: The primary outcome measure was ORR, defined as the proportion of patients with either a complete response or a partial response by investigator assessment according to RECIST v1.1.
Time Frame: 12 Months
Population: ORR was assessed on the efficacy analysis set, consisting of all patients with measurable disease, PRCC confirmed by a central laboratory and received at least 1 dose of AZD6094 (n = 85).
Measure: Count of Participants; unit: Participants
Groups:
- Total [600mg AZD6094 po]: All participants tested for the presence of c-MET mutations
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po] | Total [600mg AZD6094 po]
Number analyzed (Participants) | 37 | 40 | 8 | 85
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 3 | 0 | 0 | 3
  Stable Disease >= 5 weeks | 23 | 19 | 4 | 46
  Progression | 10 | 20 | 4 | 34
  Not Evaluable | 1 | 1 | 0 | 2

3. Primary Outcome: Objective Response Rate (RECIST Version 1.1) Stratified by c-MET Status in Safety Analysis Set
Description: The primary outcome measure was ORR, defined as the proportion of patients with either a confirmed complete response/partial response by investigator assessment according to RECIST v1.1.
Time Frame: 12 Months
Population: ORR was assessed on the safety analysis set, consisting of all patients who received at least one dose of the study drug (n = 109).
Measure: Count of Participants; unit: Participants
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po] | Total [600mg AZD6094 po]
Number analyzed (Participants) | 46 | 47 | 16 | 109
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 8 | 0 | 0 | 8
  Stable Disease >= 5 weeks | 27 | 21 | 11 | 59
  Progression | 10 | 25 | 5 | 40
  Not Evaluable | 1 | 1 | 0 | 2

4. Secondary Outcome: Progression Free Survival Stratified by c-MET Status in the Efficacy Analysis Set
Time Frame: Up to 12 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po]
Number analyzed (Participants) | 37 | 40 | 8
Weeks | 18.3 [12.3 to 35.4] | 9.7 [6.1 to 12.4] | 6.1 [5.1 to NA] — Due to insufficient number of events, the upper limit of the 95% CI for median PFS was not calculable.

5. Secondary Outcome: Overall Survival Stratified by c-MET Status in the Efficacy Analysis Set
Time Frame: Up to 12 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po]
Number analyzed (Participants) | 37 | 40 | 8
Weeks | NA [34.6 to NA] — As the sufficient number of events was not reached at the time of data cut-off, the median OS and the upper limit of the 95% CI for median OS were not calculable. | 61.1 [29.4 to NA] — Due to insufficient number of events, the upper limit of the 95% CI for median OS was not calculable. | 51.5 [8.1 to NA] — Due to insufficient number of events, the upper limit of the 95% CI for median OS was not calculable.

6. Secondary Outcome: Progression Free Survival Stratified by c-MET Status in the Safety Analysis Set
Time Frame: Up to 12 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po]
Number analyzed (Participants) | 46 | 47 | 16
Weeks | 24.7 [17.7 to 35.4] | 6.6 [6.1 to 11.9] | 12.1 [6.1 to 41.9]

7. Secondary Outcome: Overall Survival Stratified by c-MET Status in the Safety Analysis Set
Time Frame: Up to 12 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po]
Number analyzed (Participants) | 46 | 47 | 16
Weeks | NA [42.9 to NA] — As the sufficient number of events was not reached at the time of data cut-off, the median OS and the upper limit of the 95% CI for median OS were not calculable. | 61.1 [40.6 to 106.7] | 54.9 [18.4 to NA] — Due to insufficient number of events, the upper limit of the 95% CI for median OS was not calculable.

8. Secondary Outcome: Change From Baseline in Target Lesion Tumour Size at 12 Weeks in Efficacy Analysis Set
Description: 12 week summary for patients in the Efficacy analysis set, by MET status. The numbers of patients analysed represent the numbers evaluable at the 12 week timepoint.
Time Frame: 12 Weeks (at 12 weeks timepoint)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po]
Number analyzed (Participants) | 22 | 14 | 1
Percent change | -6.3 (21.56) | 3.4 (20.05) | 7.1 (0)

9. Secondary Outcome: Change From Baseline in Target Lesion Tumour Size at 12 Weeks in Safety Analysis Set.
Description: 12 week summary for patients in the Safety analysis set by MET Status. The number of patients analysed represent the number of evaluable patients at the 12 week timepoint.
Time Frame: 12 Weeks (at 12 week timepoint)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | c-MET Positive [600mg AZD6094 po] | c-MET Negative [600mg AZD6094 po] | c-MET Status Unknown [600mg AZD6094 po]
Number analyzed (Participants) | 30 | 16 | 6
Percent change | -10.9 (21.39) | 4.3 (18.96) | 5.1 (17.41)

10. Secondary Outcome: Duration of Response
Description: Duration of Response is the time from the first documentation of confirmed complete response/partial response until the date of progression, or death in the absence of progression. There were 8 responders: one of whom subsequently progressed or died and seven of whom were still classified as responders at the time of data cut-off and were therefore censored. It was not possible to determine a median or 75th percentile.
Time Frame: Up to 12 months
Measure: Median (Inter-Quartile Range); unit: Weeks
Groups:
- Safety Analysis Set [600mg AZD6094 po]: All patients who have received at least 1 dose of study medication
Arm/Group | Safety Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 109
Weeks | NA [18.1 to NA] — The median DoR and 75th percentile for DoR were not calculable within the timeframe of this study.

11. Secondary Outcome: Peak Plasma Concentration of AZD6094 Following Single Dose
Description: The number of patients analysed represent the number of patients with evaluable PK parameters for this endpoint.
Time Frame: 24 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Pharmacokinetic Analysis Set [600mg AZD6094 po]: All patients that received at least one dose of study medication and had evaluable PK data
Arm/Group | Pharmacokinetic Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 53
ng/mL | 3038.8984 (44.4184)

12. Secondary Outcome: Time to Peak Plasma Concentration of AZD6094 After Single Dose
Description: The number of patients analysed represent the number of patients with evaluable PK parameters for this endpoint.
Time Frame: 24 Hours
Measure: Median (Full Range); unit: Hours
Arm/Group | Pharmacokinetic Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 53
Hours | 2.0 [0.5 to 8.0]

13. Secondary Outcome: Apparent Volume of Distribution of AZD6094 Following Single Dose
Description: The number of patients analysed represent the number of patients with evaluable PK parameters for this endpoint.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Pharmacokinetic Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 19
Liters | 137.4237 (36.5971)

14. Secondary Outcome: Area Under Plasma Concentration Time Curve for AZD6094 After Single Dose
Description: The number of patients analysed represent the number of patients with evaluable PK parameters for this endpoint.
Time Frame: 24 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pharmacokinetic Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 19
h*ng/mL | 13144.7381 (36.4328)

15. Secondary Outcome: Area Under Plasma Concentration Time Curve for AZD6094 After Single Dose (Time Zero to Last Measurement)
Description: The number of patients analysed represent the number of patients with evaluable PK parameters for this endpoint.
Time Frame: 24 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pharmacokinetic Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 53
h*ng/mL | 13214.2441 (46.4616)

16. Secondary Outcome: Apparent Total Clearance of AZD6094 From Plasma After Single Dose
Description: The number of patients analysed represent the number of patients with evaluable PK parameters for this endpoint.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Pharmacokinetic Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 19
L/hour | 48.4938 (17.3386)

17. Secondary Outcome: Mean Residence Time of AZD6094 After Single Dose
Description: The number of patients analysed represent the number of evaluable PK parameters for this endpoint.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pharmacokinetic Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 19
Hours | 3.9837 (0.4813)

18. Secondary Outcome: Elimination Half-Life of AZD6094 After Single Dose
Description: The number of patients analysed represent the number of patients with evaluable PK parameters for this endpoint.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pharmacokinetic Analysis Set [600mg AZD6094 po]
Number analyzed (Participants) | 19
Hours | 2.0499 (0.3820)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Groups:
- AZD6094 600 mg Per Day Orally: All patients who received at least one dose of study medication
Arm/Group | AZD6094 600 mg Per Day Orally
All-Cause Mortality (participants affected / at risk) | 57/109
Serious Adverse Events (participants affected / at risk) | 27/109
Other Adverse Events (participants affected / at risk) | 107/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD6094 600 mg Per Day Orally (N=109)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Adrenal insufficiency (Endocrine disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Cellulitis (Infections and infestations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lung Infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Transaminases increased (Investigations) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Wound infection (Infections and infestations) | 1
Drug-induced Liver Injury (Hepatobiliary disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Loss of Consciousness (Nervous system disorders) | 1
Oedema (General disorders) | 1
Myocardial Infaction (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusional state (Psychiatric disorders) | 1
Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD6094 600 mg Per Day Orally (N=109)
Anaemia (Blood and lymphatic system disorders) | 17
Nausea (Gastrointestinal disorders) | 56
Vomiting (Gastrointestinal disorders) | 34
Constipation (Gastrointestinal disorders) | 29
Diarrhoea (Gastrointestinal disorders) | 18
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal distension (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 49
Peripheral oedema (General disorders) | 35
Asthenia (General disorders) | 8
Oedema (General disorders) | 8
Chest pain (General disorders) | 7
Mucosal inflammation (General disorders) | 6
Blood creatinine increased (Investigations) | 18
Aspartate aminotransferase increased (Investigations) | 15
Weight decreased (Investigations) | 14
Alanine aminotransferase increased (Investigations) | 12
Weight increased (Investigations) | 8
Blood alklaine phosphatase increased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 25
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 16
Arthalgia (Musculoskeletal and connective tissue disorders) | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Flank pain (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 8
Proteinuria (Renal and urinary disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Muscle spasm (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pain (General disorders) | 5
Chills (General disorders) | 5
Pyrexia (General disorders) | 5
Fluid retention (Metabolism and nutrition disorders) | 5
Ascites (Gastrointestinal disorders) | 5
Insomnia (Psychiatric disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 5

LIMITATIONS AND CAVEATS:
For the secondary outcome measure Duration of Response the median was not calculable because at data cut-off some participants were still responding.

Point to note: All patients on this trial received 600mg AZD6094 po.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No